CLINICAL TRIAL: NCT06686069
Title: Effect of Oral L-arginine 3.32 g a Day on Oxidative Stress Influencing Beta Cell Function and Insulin Resistance. A Phase 3, Randomized, Double-blind, Placebo-controlled Explorative Study in Overweight and Obese Patients With Pre-diabetes.
Brief Title: Effect of Oral L-arginine 3.32 g a Day on Oxidative Stress Influencing Beta Cell Function and Insulin Resistance.
Acronym: L-BIOARG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Barbara Maglione, Head of Research and Development, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 180893; 1893 (Other: San raffaele hospital)
Record Dates: First submitted 2024-11-05; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Diabetes; Pre-diabetes; Metabolic Syndrome
Keywords: L-bioarginine
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Treatment with L-arginine vs placebo
Who Masked: Participant, Investigator
Masking Description: A and B vials given by physicians to the enrolled patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo, untreated (Placebo Comparator): No treatment
  Interventions: Dietary Supplement: bioarginina zero; Dietary Supplement: Placebo
- bioarginina zero (Active Comparator): L-arginine treatment
  Interventions: Dietary Supplement: bioarginina zero; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: bioarginina zero — treatment
Dietary Supplement: Placebo — absence of treatment

SUMMARY:
The objective of this clinical trial is to explore whether L-arginine supplementation with 3.32g/day may enhance antioxidant defenses in overweight and obese patients with pre-diabetes and metabolic syndrome, possibly providing beta cell function and insulin resistance improvement. The primary efficacy endpoint will be to explore the effects of a short-term L-arginine supplementation on AOPP levels and PAI after three months of treatment, based on the rationale explained above. Secondary, the effects of L-arginine supplementation on lipid peroxidation products and antioxidant defenses will be explored. Tertiary, the effects of L-arginine supplementation on insulin resistance and glucose metabolism parameters will be also evaluated.

DETAILED DESCRIPTION:
Recent studies have demonstrated beneficial effects of the use of L-arginine supplementation as a nutrient treatment in diabetes and prediabetes, with documented beneficial effects on β- cell function and insulin sensitivity .

A long-term follow-up randomized clinical trial also demonstrated a reduced cumulative incidence of type 2 diabetes among subjects at high risk of developing the disease . The same study reported a significantly AOPP levels reduction at 18 months in L-arginine arm compared to placebo and this effect was maintained through the 108 months of follow up. Indeed, AOPP levels decreased by 26.1% at 18 months, remaining lower during the post intervention period in L-arginine group.

However, in this study, AOPP levels were firstly evaluated at baseline and then only 18 months after starting treatment. Therefore, to date, no data are currently available regarding the effects of a short-term treatment on AOPPs levels. In addition, data in vivo on rats suggest a rapid improvement in antioxidant defense and in total antioxidative capacity in plasma and liver after a 14 days treatment period with L-arginine.

Advanced oxidation protein products are formed during oxidative stress by myeloperoxidase action in activated neutrophils through chloraminated oxidants production. AOPPs molecular structure is similar to advanced glycation endproducts (AGEs) as they have similar biological activities. Precisely, AOPPs exert induction of proinflammatory cytokines and adhesion molecules maintaining inflammatory pathways activated and favoring pro-oxidant state. In addition, many reports highlighted a strict correlation between AOPPs and glucose metabolism suggesting being an early marker of diabetes mellitus and metabolic syndrome. The prooxidant-antioxidant index (PAI) has been proposed as possible marker of MetS. It is expressed as the ratio between the AOPP levels and the total radical-trapping antioxidant capacity (TRAP), a surrogate for the total antioxidant defenses in the plasma. An interesting study by Venturini et al. evidenced the relationship between AOPPs and MetS also highlighting that PAI progressively increased (P <0.05) according to the number of MetS components, whereas AOPPs and total radical-trapping antioxidant parameter increased (P <0.05) when 5 components were compared with 3 and 4 components .

Lipid peroxidation products such as malondialdehyde (MDA), and 4-hydroxynonenal (HNE) have been reported to be highly related to inflammation and MetS. These molecules are considered important biomarkers of oxidative stress because of the high susceptibility of polyunsaturated fatty acids-rich cell membranes to lipid peroxidation when exposed to ROS or other free radicals . A positive correlation has been described by several studies among obesity, IR, MetS, glycaemic control and MDA and HNE levels.

Regarding the antioxidant enzymes, a study by Lang et al. on rats fed with L-arginine for 14 days demonstrated a significant stimulation in GSH synthesis enzymes, CAT, SOD and GPx activity and mRNA expression enhancing the total antioxidative capacity in plasma (T-AOC or TRAP) and in the liver strongly suggesting that L-arginine oral administration can ameliorate antioxidant defenses.

To conduct this study, the investigators selected a L-arginine dosage of 3,32 g/day, based on evidence that this dosage was associated to an improvement of the inflammatory response and beneficial modulating of oxidative stress in favor of an antioxidant state.

ELIGIBILITY:
Inclusion Criteria:

* consented male and female patients aged 20-70 years with Body Mass Index (BMI) >25 kg/m2,
* pre-diabetes (fasting glucose 100-125 mg/dL and HbA1c 5.7-6.5%) or metabolic syndrome, defined according to modified NCEP-ATP III criteria (Grundy SM et al., Circulation, 2005) as the presence of three or more of the following clinical features: blood glucose levels >100 mg/dL, HDL-cholesterol <40 mg/dL in males and <50 mg/dL in females, triglycerides levels >150 mg/dL, waist circumference >102 cm in males and >88 cm in females and hypertension, defined as repeated blood pressure measurements >130/85 mmHg.

Exclusion Criteria:

* moderate to severe renal impairment (calculated creatinine clearance (CrCl) <60 mL/min according to the Cockcroft-Gault formula);
* hepatic dysfunction (ALT/AST >3 x upper limit of normal and total bilirubin >3 mg/dL);
* hypoalbuminemia (serum albumin <3 g/dL);
* history of any past or current clinically significant cardiovascular diseases;
* monogenic, secondary and pharmacological causes of diabetes and obesity;
* any other clinical condition/disease that the Principal Investigator believes might confound study outcome;
* patients on treatment with insulin or any anti-diabetic drugs or medications known to influence glucose tolerance will also be excluded;
* pregnant or breast-feeding women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-01-18 (Estimated); Primary Completion 2025-11-18 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
effects of a short-term L-arginine supplementation on AOPP levels after three months of treatment | 3 months
  effects of a short-term L-arginine supplementation on AOPP levels and PAI after three months of treatment

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT06686069/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT06686069/ICF_001.pdf